CLINICAL TRIAL: NCT03046303
Title: Radical Gastrectomy Within Enhanced Recovery Programs: a Prospective Randomized Controlled Trial
Brief Title: Radical Gastrectomy Within Enhanced Recovery Programs(ERAS): a Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS for Radical gastrectomy
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Gastrostomy Complications
Keywords: ERAS,gastric cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Patients were admitted 1-3 days prior to their respective dates of operation. A ERAS protocol was used in the ERAS group.
  Interventions: Procedure: ERAS
- conventional pathway group (No Intervention): The conventional pathway group received conventional care.

INTERVENTIONS:
Procedure: ERAS — optimized pain control, restricted I.V. fluids, early initiation of post-operative oral feeding and enforced mobilization
  Arms: ERAS group

SUMMARY:
This study is a prospective, single-center, randomized controlled trial. The study protocol was approved by the Ethics Committee at the First Hospital of Jilin University.ERAS is combined with the laprascopic gastrectomy to assess the efficacy and safety in patients with advanced gastric carcinoma.The hospitalized patients were randomly divided into ERAS group and conventional pathway group . Inter-group differences were evaluated for clinical recovery index, economic indicators, length of hospital stay, 3 years to 5 years long-term survival, etc.

ELIGIBILITY:
Inclusion Criteria:

* (1) A preoperative cancer stage of T2, T3, T4, Any N, M0 without digestive obstruction confirmed by whole body CT scan, which could be treated with laparoscopic gastrectomy; (2) age 18-75 years; (3) pathologic confirmation of gastric adenocarcinoma by endoscopic biopsy; (4) normal hematological, renal, hepatic, and cardiac parameters, ASA score < III without severe systemic disease; and (5) no history of treatment with neoadjuvant chemotherapy and/or radiotherapy.

Exclusion Criteria:

* patients requiring conversion to open gastrectomy; excessive bleeding (˃ 500 mL);and patients opting out of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
clinical parameters | One week after operation
  length of post-operative stay

SECONDARY OUTCOMES:
Postoperative complications | 30 days after operation
  wound infection;post-opeartion bleeding;ileus;stenosis;leakage

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No